CLINICAL TRIAL: NCT01941394
Title: Pilot Study for Safety and Effectiveness Assessment of Bone Marrow Mesenchymal Stem Cell Infusion for Acute Graft-versus-host Disease Prophylaxis and Treatment After Allogenic Bone Marrow Transplantation
Brief Title: Mesenchymal Stem Cells Infusion for aGVHD Prophylaxis Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, Head of BMT department, National Research Center for Hematology, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NRCH-MSC
Record Dates: First submitted 2013-08-30; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Graft-versus-host Disease; Relapse
Keywords: GVHD; Relapse; Overall Survival
MeSH Terms: conditions — Graft vs Host Disease; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With MSC (Experimental): infusion of Mesenchymal stem cells at dose 1 mln cells per kg
  Interventions: Biological: Mesenchymal stem cells
- Without MSC (No Intervention): Without MSC infusion

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cells infusion
  Other Names: Mesenchymal stem cells infusion
  Arms: With MSC

SUMMARY:
Infusion of Mesenchymal Stem Cell (MSC) at day of recovery after bone marrow transplant (BMT) for patients with AL, AA and MM for acute Graft-versus-host Disease (GVHD) prophylaxis and treatment.

DETAILED DESCRIPTION:
Infusion of mesenchymal stem cells at day of recovery after BMT for patients with AL, AA and MM for acute GVHD prophylaxis and treatment. Infusion at dose 1 cells mln/kg at day of white blood cells recovery.

ELIGIBILITY:
Inclusion Criteria:

* allogenic BMT from related or unrelated donor

Exclusion Criteria:

* Severe infection
* Relapse
* admission to ICU
* refusal of research
* patients with graft failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
GVHD | Every 30 day for 1 year after BMT

SECONDARY OUTCOMES:
Overall survival | Every 30 day for 1 year after BMT
Relapse-free survival | Every 30 day for 1 year after BMT
Infection rate | Every 30 day for 1 year after BMT

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parovichnikova, Prof MD PhD, Principal Investigator — National Research Center for Hematology
Locations (1):
- BMT department, Moscow, Russia

REFERENCES:
- [Result] Kuzmina LA, Petinati NA, Parovichnikova EN, Lubimova LS, Gribanova EO, Gaponova TV, Shipounova IN, Zhironkina OA, Bigildeev AE, Svinareva DA, Drize NJ, Savchenko VG. Multipotent Mesenchymal Stromal Cells for the Prophylaxis of Acute Graft-versus-Host Disease-A Phase II Study. Stem Cells Int. 2012;2012:968213. doi: 10.1155/2012/968213. Epub 2011 Dec 25. PMID 22242033
- [Derived] Petinati N, Davydova Y, Nikiforova K, Bigildeev A, Belyavsky A, Arapidi G, Drize N, Kuzmina L, Parovichnikova E, Savchenko V. T Cell and Cytokine Dynamics in the Blood of Patients after Hematopoietic Stem Cell Transplantation and Multipotent Mesenchymal Stromal Cell Administration. Transplant Cell Ther. 2023 Feb;29(2):109.e1-109.e10. doi: 10.1016/j.jtct.2022.10.030. Epub 2022 Nov 11. PMID 36372356